CLINICAL TRIAL: NCT01283581
Title: A Phase 2 Exploratory Study of Objective Endpoints in Subjects With Acute Bacterial Skin and Skin Structure Infections Treated With Delafloxacin, Vancomycin, or Linezolid
Brief Title: A Study to Assess Objective Endpoint Measurements of Response in Bacterial Skin Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RX-3341-202
Record Dates: First submitted 2011-01-24; First posted 2011-01-26 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Skin and Subcutaneous Tissue Bacterial Infections
MeSH Terms: interventions — delafloxacin; Linezolid; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Delafloxacin (Experimental): 300 mg IV (intravenous) every 12 hours for 5-14 days
  Interventions: Drug: Delafloxacin
- Vancomycin (Active Comparator): 15 mg/kg, up to 1250 mg, IV every 12 hours for 5-14 dyas
  Interventions: Drug: Vancomycin
- Linezolid (Active Comparator): 600 mg IV every 12 hours for 5-14 days
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Delafloxacin — 300mg IV every 12 hours for 5-14 days
  Other Names: RX-3341
  Arms: Delafloxacin
Drug: Linezolid — 600mg IV every 12 hours for 5-14 days
  Other Names: Zyvox
  Arms: Linezolid
Drug: Vancomycin — 15mg/kg, up to 1250 mg, IV every 12 hours for 5-14 days
  Other Names: Vancocin
  Arms: Vancomycin

SUMMARY:
The purpose of this study is to compare clinical response to the measurement techniques of several objective measures of clinical efficacy for use in future ABSSSI (Acute Bacterial Skin and Skin Structure Infection) clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years of age) men or women
* Sexually active women and men with partners of childbearing potential must agree to use an acceptable form of contraception as determined by the investigator during participation in the study and for 30 days after the final dose of study drug
* Female partners of male subjects should also use an additional reliable method of contraception during study and for 30 days after the final dose of study drug
* Subjects must have a diagnosis of ABSSSI - one or more of the following 4 infection types: cellulitis/erysipelas, wound infection, major cutaneous abscess, or burn infection
* Subjects must have lymph node enlargement due to the present infection or at least one of the following symptoms of systemic infection: fever ≥ 38°C, lymphangitis, WBC (white blood cell) count ≥ 15,000 cells/μL, elevated C-reactive protein (> 5.0mg/L)
* In the opinion of the investigator, the subject must require and be a suitable candidate for IV antibiotic therapy

Exclusion Criteria:

* A medical history of significant hypersensitivity or allergic reaction to quinolones, linezolid, vancomycin, or vancomycin derivatives
* Women who are pregnant or lactating
* Any chronic or underlying skin condition at the site of infection that may complicate the assessment of response
* Subjects with any of the following: infection involving prosthetic materials or foreign bodies, infection associated with a human or animal bite, osteomyelitis, decubitus ulcer, diabetic foot ulcer, septic arthritis, mediastinitis, necrotizing fasciitis, anaerobic cellulitis, or synergistic necrotizing cellulitis, myositis, tendinitis, endocarditis, toxic shock syndrome, gangrene, burns covering ≥ 10% of body surface area, severely impaired arterial blood supply, current evidence of deep vein thrombosis or superficial thrombophlebitis
* Minor abscesses, unless present with one of the ABSSSI types
* Any infection expected to require other antimicrobial agents in addition to study drug
* Receipt of > 24 hours of systemic antibiotic therapy in the 14 days before enrollment unless one of the following is documented: the subject received a single dose of a short-acting antibacterial drug 3 or more days before clinical trial enrollment for surgical prophylaxis or recently completed treatment with an antibacterial drug for an infection other than ABSSSI and the drug does not have antibacterial activity against bacterial pathogens that cause ABSSSI
* Receipt of more than 1 dose of a potentially effective antibacterial agent for treatment of the ABSSSI under study prior to enrollment
* Receipt of chronic anti-inflammatory therapy for longer than 14 days before enrollment
* Severely compromised immune systems
* Subjects taking any medicinal product which inhibits monoamine oxidases A or B or within 2 weeks of Screening
* Hypertension as defined by a systolic blood pressure of ≥ 180 mmHg or a diastolic blood pressure of ≥110 mmHg with confirmed re-check within 20 minutes of initial reading
* Subjects with pheochromocytoma, thyrotoxicosis and/or subjects taking any of the following types of medications: sympathomimetic agents, vasopressive agents, dopaminergic agents, or other agents with the potential for serotonergic interactions
* Subjects with carcinoid syndrome and/or subjects taking any of the following medications: serotonin re-uptake inhibitors, tricyclic antidepressants, serotonin 5-HT1 (serotonin receptor) receptor agonists, meperidine, or buspirone
* Known history of liver disease
* History of severe renal impairment
* Life expectancy of < 3 months
* Any underlying disease that, in the opinion of the investigator, could interfere with the subject's ability to participate in the study
* Subjects previously randomized in this study or in who have received a dose of an investigational drug within 30 days of randomization
* Subjects > 140 kg in body weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hopkins, MD, Study Director
Locations (31):
- United States (31):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Drug Research and Analysis Corp, Montgomery, Alabama
  - Southbay Pharma Research, Buena Park, California
  - eStudySite, Chula Vista, California
  - eStudySite, La Mesa, California
  - HealthCare Partners Medical Group, Los Angeles, California
  - eStudySite, Oceanside, California
  - HealthCare Partners Medical Group, Pasadena, California
  - Christiana Care Health Services, Newark, Delaware
  - Riverside Clinical Research, Edgewater, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Central Florida Internists, Kissimmee, Florida
  - Central Florida Internists Medical, Orlando, Florida
  - Central Florida Internists, Saint Cloud, Florida
  - Ronald Barbour, MD, Temple Terrace, Florida
  - Southeast Regional Research Group, Columbus, Georgia
  - Atlanta Institute for Medical Research, Inc, Decatur, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Four Rivers Clinical Research, Inc, Paducah, Kentucky
  - Medical Development Centers, LLC, Baton Rouge, Louisiana
  - University of Missouri Health Care, Columbia, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - eStudySite, Las Vegas, Nevada
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Remington-Davis, Inc., Columbus, Ohio
  - Ravi Kamepalli, MD, Lima, Ohio
  - Health Concepts, Rapid City, South Dakota
  - Jennifer Johnson-Caldwell, MD, Houston, Texas
  - Alan Nolasco, MD, Houston, Texas

REFERENCES:
- [Result] Results of a Phase 2 Study of Delafloxacin (DLX) Compared to Vancomycin (VAN) and Linezolid (LNZ) in Acute Bacterial Skin and Skin Structure Infections (ABSSSI) J. Longcor 1 , S. Hopkins 1 , L. Lawrence 1 , S. Green 2 , P. Mehra 2 , P. Manos 2 , W. Sears 2 , W. O'Riordan 2 1 Rib - X Pharmaceuticals, Inc., New Haven, CT; 2 eStudySite, San Diego, CA 52nd ICAAC, San Francisco, CA 2012
- [Result] Characterization and In Vitro Activity of Delafloxacin (DLX) Against Isolates from a Phase 2 Study of Acute Bacterial Skin and Skin Structure Infections (ABSSSI) L. Lawrence 1 , S. Hopkins 1 , D. Sahm 2 , Jennifer Deane 2 , E. Burak 1 , J. Longcor 1 1 Rib - X Pharmaceuticals, Inc., New Haven, CT; 2 Eurofins Medinet, Chantilly, VA 52nd ICAAC, San Franciso, 2012
- [Result] Pharmacokinetics (PK) of Delafloxacin (DLX), Vancomycin (VAN), and Linezolid (LNZ) in a Phase 2 Exploratory Study in Subjects with Acute Bacterial Skin and Skin Structure Infections (ABSSSI) R. Hoover 1 , L. Lawrence 1 , J. Longcor 1 , J. Greenfield 2 1 Rib - X Pharmaceuticals, New Haven, CT; 2 PharmaNet/i3, The Woodlands, TX 52nd ICAAC, San Francisco, CA, 2012
- [Derived] Kingsley J, Mehra P, Lawrence LE, Henry E, Duffy E, Cammarata SK, Pullman J. A randomized, double-blind, Phase 2 study to evaluate subjective and objective outcomes in patients with acute bacterial skin and skin structure infections treated with delafloxacin, linezolid or vancomycin. J Antimicrob Chemother. 2016 Mar;71(3):821-9. doi: 10.1093/jac/dkv411. Epub 2015 Dec 17. PMID 26679243

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study targeted patients with ABSSSI (acute bacterial skin and skin structure infections), defined as cellulitis/erysipelas, wound infection, major cutaneous abscess, or burn infection; the minimum surface area was to be 75 square centimeters.
Groups:
- Delafloxacin IV (Intravenous): Delafloxacin 300 mg, BID (twice a day)
- Linezolid IV: Linezolid 600 mg, BID
- Vancomycin IV: Vancomycin 15 mg/kg or up to 1250 mg/dose, BID
Period: Overall Study
Arm/Group | Delafloxacin IV (Intravenous) | Linezolid IV | Vancomycin IV
Started | 81 | 77 | 98
Completed | 69 | 63 | 78
Not Completed | 12 | 14 | 20
Not completed — Lost to Follow-up | 8 | 6 | 8
Not completed — Withdrawal by Subject | 2 | 5 | 2
Not completed — Adverse Event | 1 | 1 | 4
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Noncompliance | 1 | 0 | 0
Not completed — Investigator unblinded | 0 | 0 | 1
Not completed — "Early termination" | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT (intent-to-treat) population, defined as all subjects who were randomized.
Groups:
- Linezolid: Linezolid 600 mg, BID
- Vancomycin: Vancomycin 15 mg/kg or up to 1250 mg/dose, BID
- Total: Total of all reporting groups
Arm/Group | Delafloxacin IV (Intravenous) | Linezolid | Vancomycin | Total
Number analyzed (Participants) | 81 | 77 | 98 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (14.26) | 44.8 (14.91) | 44.8 (15.54) | 43.2 (15.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 25 | 47 | 104
  Male | 49 | 52 | 51 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 11 | 27 | 57
  Not Hispanic or Latino | 62 | 66 | 71 | 199
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 2 | 7
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 3
  Black or African American | 10 | 15 | 15 | 40
  White | 63 | 58 | 74 | 195
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 4 | 7
Baseline Infection Category [Number; unit: Participants] — Categories of infection included major cutaneous abscess, cellulitis/erysipelas, wound infection, or burn infection
  Participants
    Major cutaneous abscess | 22 | 24 | 29 | 75
    Cellulitis/erysipelas | 38 | 31 | 44 | 113
    Wound infection | 19 | 20 | 23 | 62
    Burn infection | 2 | 2 | 1 | 5
    Not assessed | 0 | 0 | 1 | 1
Pathogens isolated at baseline [Number; unit: Participants]
  Subjects with at least 1 pathogen | 51 | 57 | 67 | 175
  Subjects with multiple pathogens | 6 | 15 | 8 | 29
  Subjects with positive blood cultures | 0 | 6 | 1 | 7
  Subjects without pathogens | 30 | 20 | 31 | 81
  Subjects with at least 1 Staphylococcus aureus | 45 | 53 | 61 | 159
  Subjects with at least 1 MRSA | 34 | 37 | 35 | 106
  Subjects with at least 1 MSSA | 11 | 16 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Assessment of Clinical Response in the ITT (Intent-to-treat) Population at Follow-up
Description: The primary efficacy endpoint was the success rate, defined as (cure)/(cure + failure), and expressed as a percentage. Cure was defined as the complete resolution of all baseline signs and symptoms of ABSSSI and follow-up and late follow-up. If erythema was the only sign of infection present at follow-up and it was then absent at late follow-up, the case was classified as a Cure.
Time Frame: Follow-up (Day 14 ± 1)
Population: ITT (intent-to-treat) population, defined as all subjects who were randomized.
Measure: Number; unit: Participants
Groups:
- Delafloxacin IV: Delafloxacin 300 mg, BID
Arm/Group | Delafloxacin IV | Linezolid | Vancomycin
Number analyzed (Participants) | 81 | 77 | 98
Participants | 57 | 50 | 53

2. Secondary Outcome: Erythema Clinical Success
Description: The number of ITT subjects who had cessation of erythema within 48-72 hours, based on digital measurements, as well as resolution/absence of fever. Cessation was defined as a percentage change from baseline in total area of erythema/induration that is less than or equal to 0%.
Time Frame: 48 - 72 hours
Population: ITT (intent-to-treat) population, defined as all subjects who were randomized.
Measure: Number; unit: Participants
Arm/Group | Delafloxacin IV | Linezolid | Vancomycin
Number analyzed (Participants) | 81 | 77 | 98
Participants | 61 | 56 | 69

3. Secondary Outcome: Pharmacokinetic (PK) Parameter, Area Under Curve, (AUCinf, ug*h/mL), in Subjects Administered Delafloxacin, Vancomycin, and Linezolid
Description: Blood samples for pharmacokinetic analyses were drawn from all subjects on Day 3 (± 1 day) of treatment within 2 hours before the first study drug infusion and at 1, 2, 3, 5, and 12 hours (ie, immediately before the second dose) after the start of the first study drug infusion. An analytical, validated method was used to analyze samples and determine human plasma concentrations. The primary pharmacokinetic parameter calculated was area under the plasma concentration - time curve from time 0 extrapolated to infinity (AUCinf, ug*h/mL).
Time Frame: Through Day 3 (± 1 day)
Population: AUCinf (ug*h/mL) for delafloxacin, linezolid, and vancomycin are presented only for those subjects with PK samples collected.
Measure: Mean (Standard Deviation); unit: ug*h/mL
Groups:
- Delafloxacin: 300 mg IV every 12 hours for 5-14 days
  Delafloxacin: 300mg IV every 12 hours for 5-14 days
Arm/Group | Delafloxacin | Vancomycin | Linezolid
Number analyzed (Participants) | 57 | 35 | 42
ug*h/mL | 23.4 (11.70) | 266.8 (88.63) | 106.0 (47.33)

4. Secondary Outcome: The Levels of Inflammation Were Examined by Measuring a Surrogate, C-Reactive Protein (CRP)
Description: CRP Levels (g/m3) were analyzed from blood samples collected from subjects at Baseline and various time points throughout the study. Change in baseline values were analyzed using an analysis of covariance (ANCOVA) model with treatment, infection category, and prior antimicrobial therapy as fixed effects and the baseline measure as the covariate.
Time Frame: Baseline, Days 1, 5, Follow-up (FU), and late Follow-up (LFU)
Population: Only subjects from ITT population with CRP levels evaluated were included in outcome measure analysis.
Measure: Mean (Standard Deviation); unit: g/m3
Arm/Group | Delafloxacin | Vancomycin | Linezolid
Number analyzed (Participants) | 81 | 98 | 77
g/m3
  Baseline: number analyzed (Participants) | 71 | 92 | 71
  Baseline | 46.6 (70.66) | 55.2 (69.70) | 49.3 (56.14)
  Day 1: number analyzed (Participants) | 70 | 90 | 68
  Day 1 | 44.2 (67.63) | 49.6 (58.56) | 49.8 (61.66)
  Day 5: number analyzed (Participants) | 76 | 94 | 72
  Day 5 | 19.6 (35.97) | 19.5 (22.63) | 26.5 (48.44)
  FU: number analyzed (Participants) | 77 | 94 | 72
  FU | 9.4 (17.65) | 11.9 (28.71) | 12.1 (26.04)
  LFU: number analyzed (Participants) | 77 | 94 | 72
  LFU | 10.8 (17.47) | 9.3 (16.46) | 12.6 (27.10)

5. Secondary Outcome: Microbiological Response Rate in All Subjects (Microbiological Evaluable Population)
Description: Based on the results of the baseline and follow up cultures and susceptibility testing, together with the clinical response assigned by the investigator, the sponsor determined a microbiological response for subjects in the ME population.
Time Frame: Follow-up (Day 14 ± 1)
Population: Microbiologically Evaluable (ME) Population - All Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Vancomycin | Linezolid
Number analyzed (Participants) | 34 | 52 | 39
Participants
  Documented Eradicated | 0 | 0 | 0
  Presumed Eradicated | 30 | 42 | 32
  Documented Persisted | 0 | 0 | 1
  Presumed Persisted | 4 | 10 | 6

6. Secondary Outcome: Microbiological Response Rate in Subjects With MRSA (Methicillin Resistant Staphylococcus Aureus) in Microbiological Evaluable (ME) Population
Description: as for outcome 5
Time Frame: Follow-up (Day 14 ± 1)
Population: Microbiologically Evaluable (ME) Population - MRSA Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Vancomycin | Linezolid
Number analyzed (Participants) | 21 | 26 | 25
Participants
  Documented Eradicated | 0 | 0 | 0
  Presumed Eradicated | 18 | 23 | 20
  Documented Persisted | 0 | 0 | 1
  Presumed Persisted | 3 | 3 | 4

7. Secondary Outcome: Clinical Response in Subjects With Infections Caused by MRSA - Microbiological ITT (MITT) Population
Description: The success rate, defined as (cure)/(cure + failure), and expressed as a percentage. Cure was defined as the complete resolution of all baseline signs and symptoms of ABSSSI and follow-up and late follow-up. If erythema was the only sign of infection present at follow-up and it was then absent at late follow-up, the case was classified as a Cure.
Time Frame: Follow-up (Day 14 ± 1)
Population: Microbiological ITT Population (MITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Vancomycin | Linezolid
Number analyzed (Participants) | 29 | 32 | 34
Participants | 19 | 21 | 21

ADVERSE EVENTS:
Description: The safety population in this study was defined as all enrolled subjects who received at least 1 dose of study drug. The respective subjects numbers were 78 (delafloxacin), 75 (linezolid), and 96 (vancomycin).
Arm/Group | Delafloxacin IV | Linezolid | Vancomycin
Serious Adverse Events (participants affected / at risk) | 5/78 | 2/75 | 6/96
Other Adverse Events (participants affected / at risk) | 59/78 | 54/75 | 62/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin IV (N=78) | Linezolid (N=75) | Vancomycin (N=96)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delafloxacin IV (N=78) | Linezolid (N=75) | Vancomycin (N=96)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 5 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 17 (17) | 16 (16) | 13 (13)
Vomiting (Gastrointestinal disorders) | 10 (10) | 6 (6) | 8 (8)
Fatigue (General disorders) | 5 (5) | 3 (3) | 6 (6)
Infusion Site Pain (Gastrointestinal disorders) | 4 (4) | 7 (7) | 5 (5)
Abscess Limb (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3) | 3 (3) | 5 (5)
Skin Infection (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Vulvovaginal Mycotic Infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 5 (5) | 5 (5)
Pruritis (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6) | 20 (20)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days